CLINICAL TRIAL: NCT00891527
Title: Adjunct Targeted Biologic Inhibition in Children With Multivessel Intraluminal Pulmonary Vein Stenosis
Brief Title: Pilot Study Using Avastin and Gleevec to Treat the Progression of Intraluminal Pulmonary Vein Stenosis
Acronym: PVS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Kathy Jenkins, Kathy J. Jenkins, MD, MPH, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07060249
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Results first posted 2017-05-31 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Pulmonary Veno Occlusive Disease
Keywords: Pulmonary Vein Stenosis,; Avastin and Gleevec,; Targeting VEGF and PDGF
MeSH Terms: conditions — Pulmonary Veno-Occlusive Disease; Stenosis, Pulmonary Vein | interventions — Bevacizumab; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Avastin and/or Gleevec (Experimental): Patients were all treated with Gleevec (imatinib mesylate) and those without congenital heart disease and those who progressed were also treated with Avastin (bevacizumab).
  Interventions: Drug: Bevacizumab (Avastin) and Imatinib Mesylate (Gleevec)

INTERVENTIONS:
Drug: Bevacizumab (Avastin) and Imatinib Mesylate (Gleevec) — Imatinib Mesylate Orange to grayish orange, opaque, 100mg capsules dissolved in 50-100mls of mineral water or apple juice. Given at 340mg/m2 once daily, preferably with a meal.
  Bevacizumab Clear to slightly opalescent liquid. Given at 10mg/kg once every 2 weeks IV. The calculated dose should be placed in an IV bag and diluted with 0.9% sodium chloride to obtain a final volume of 25-100mls. The vials contain no antibacterial preservatives. Once diluted, must be administered within 8 hrs. Initially administered over 90 mins. If no adverse reactions occur, 2nd dose administered over 60 mins. If still no adverse reactions, subsequent doses administered over 30 mins. If infusion-related adverse reactions occur, further infusions administered over the shortest period that was well tolerated.
  Other Names: Bevacizumab (rhuMAb VEGF, Avastin), NSC 704865; Imatinib Mesylate (Gleevec, STI571), NSC 716051, IND 61,135

SUMMARY:
The objective of this study is to conduct a pilot study using biologic agents Avastin and Gleevec to treat progression of multivessel intraluminal pulmonary vein stenosis in children.

DETAILED DESCRIPTION:
Intraluminal pulmonary vein stenosis is rare but life threatening disease that affects both infants and children. It can be isolated to a single pulmonary vein, but most often occurs in multiple vessels simultaneously. It can occur as a complicating feature of complex congenital heart disease, but can also occur in isolation in infants with otherwise normal hearts. Response to conventional surgical or transcatheter-based therapies is usually short-lived. Typically within 3 to 4 weeks the obstruction recurs. Repeat surgical attempts provide only temporary relief and eventually all of these infants die without lung transplantation.

While the cause of this disease is unknown the mechanism of progressive obstruction has recently been determined through biopsy and autopsy reviews to result from neo-proliferative cells identified as myofibroblasts which have cell markers VEGF and PDGF. Chemotherapeutic agents Avastin and Gleevec have shown to inhibit myo-proliferation through these markers. The overall objective of this protocol is to conduct a pilot study using the biologic agents Avastin and Gleevec to treat progression of intraluminal pulmonary vein stenosis (PVS). From this pilot group of 10 patients we will attempt to provide an enhanced characterization of the progressive primary disease process, as well as its secondary manifestations. Results will be analyzed descriptively; data gathered from this pilot study will be used to inform further study examining safety and efficacy outcomes. Initial study was limited to 10 patients, but was later expanded to 50 enrolled patients.

The study objectives will be accomplished by achievement of the following Specific Aims:

1. To describe the feasibility of administration of Gleevec® with or without Avastin® to treat the progression of intraluminal PVS in patients with multivessel disease. Patients with PVS in conjunction with congenital heart disease (CHD) will receive Gleevec® alone, with Avastin® added if significant progression occurs; patients with primary PVS and PVS in conjunction with lung disease will be treated with both drugs simultaneously.
2. To characterize the time to progression and the proportion of patients who survive 48 weeks after enrollment.
3. To describe the toxicity associated with administration of Gleevec® with or without Avastin® during a 48 week course of treatment among patients with multivessel PVS.

Patients will be treated with Gleevec® with or without Avastin® for a period of 48 weeks, and will be followed until 72 weeks. Clinical status will be assessed by serial lab testing, monthly echocardiography and lung scans, and baseline and q24 week CT angiography or angiography. Obstruction of individual pulmonary veins will be assessed using a standard score, and patients will be classified as stabilized, recurred or progressed based on changes in the individual vein scores.

ELIGIBILITY:
Eligibility Criteria: (Both groups)

* Evidence of intraluminal pulmonary vein stenosis in > 1 vessel
* Evidence of myofibroblast neo-proliferation, if biopsies were obtained
* Acceptable organ function includes:

Creatinine < 1.5 x normal for age. Bilirubin < 1.5 x normal for age. ALT < or = 5x normal ANC > or = 1,500/mm3, Hemoglobin > or = 10g/dl, Platelets > or = 100,000/mm3.

Group A Eligibility Criteria: (begin treatment with Gleevec® only)

* Significant concomitant congenital heart defect
* Disease severity for each vessel Category 5 or lower or Category 6 or 7 in no more than 1 vessel

Group B Eligibility Criteria: (begin treatment with Gleevec® and Avastin®)

* Primary PVS (i.e. without concomitant congenital heart defect or lung disease)
* Significant concomitant lung disease
* Patients with PVS and underlying CHD who have category 6 or 7 disease in at least 2 of their pulmonary veins even after surgical or cath-based interventions.
* Accepted organ function includes:

Urine protein < 1

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy J Jenkins, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Childrens Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bini RM, Cleveland DC, Ceballos R, Bargeron LM Jr, Pacifico AD, Kirklin JW. Congenital pulmonary vein stenosis. Am J Cardiol. 1984 Aug 1;54(3):369-75. doi: 10.1016/0002-9149(84)90199-1. PMID 6465018
- [Background] Webber SA, de Souza E, Patterson MW. Pulsed wave and color Doppler findings in congenital pulmonary vein stenosis. Pediatr Cardiol. 1992 Apr;13(2):112-5. doi: 10.1007/BF00798218. PMID 1614915
- [Background] Adey CK, Soto B, Shin MS. Congenital pulmonary vein stenosis: a radiographic study. Radiology. 1986 Oct;161(1):113-7. doi: 10.1148/radiology.161.1.3763853.
- [Background] Mendelsohn AM, Bove EL, Lupinetti FM, Crowley DC, Lloyd TR, Fedderly RT, Beekman RH 3rd. Intraoperative and percutaneous stenting of congenital pulmonary artery and vein stenosis. Circulation. 1993 Nov;88(5 Pt 2):II210-7. PMID 8222156
- [Background] Driscoll DJ, Hesslein PS, Mullins CE. Congenital stenosis of individual pulmonary veins: clinical spectrum and unsuccessful treatment by transvenous balloon dilation. Am J Cardiol. 1982 May;49(7):1767-72. doi: 10.1016/0002-9149(82)90257-0. PMID 6211076
- [Background] Bahl VK, Chandra S, Mishra S. Congenital stenosis of isolated pulmonary vein: role of retrograde pulmonary vein catheterization. Int J Cardiol. 1997 Jun 27;60(1):103-5. doi: 10.1016/s0167-5273(97)02972-0. PMID 9209947
- [Background] Mendeloff EN, Spray TL, Huddleston CB, Bridges ND, Canter CB, Mallory GB Jr. Lung transplantation for congenital pulmonary vein stenosis. Ann Thorac Surg. 1995 Oct;60(4):903-6; discussion 907. doi: 10.1016/0003-4975(95)00543-t. PMID 7574992
- [Background] Martinez-Climent J, Cavalle T, Ferris Tortajada J. Non-malignant tumors that can mimic cancer during the neonatal period. Eur J Pediatr Surg. 1995 Jun;5(3):156-9. doi: 10.1055/s-2008-1066193. PMID 7547802
- [Background] Herman TE, Siegel MJ. Special imaging casebook. Infantile myofibromatosis: solitary and multifocal varieties. J Perinatol. 1995 May-Jun;15(3):250-2. No abstract available. PMID 7666279
- [Background] Davies RS, Carty H, Pierro A. Infantile myofibromatosis--a review. Br J Radiol. 1994 Jul;67(799):619-23. doi: 10.1259/0007-1285-67-799-619. PMID 8061994
- [Background] Hutchinson L, Sismanis A, Ward J, Price L. Infantile myofibromatosis of the temporal bone: a case report. Am J Otol. 1991 Jan;12(1):64-6. PMID 2012194
- [Background] Goldberg NS, Bauer BS, Kraus H, Crussi FG, Esterly NB. Infantile myofibromatosis: a review of clinicopathology with perspectives on new treatment choices. Pediatr Dermatol. 1988 Feb;5(1):37-46. doi: 10.1111/j.1525-1470.1988.tb00882.x. PMID 3288983
- [Background] Duffy MT, Harris M, Hornblass A. Infantile myofibromatosis of orbital bone. A case report with computed tomography, magnetic resonance imaging, and histologic findings. Ophthalmology. 1997 Sep;104(9):1471-4. doi: 10.1016/s0161-6420(97)30114-6. PMID 9307643
- [Background] Coffin CM, Neilson KA, Ingels S, Frank-Gerszberg R, Dehner LP. Congenital generalized myofibromatosis: a disseminated angiocentric myofibromatosis. Pediatr Pathol Lab Med. 1995 Jul-Aug;15(4):571-87. doi: 10.3109/15513819509026993. PMID 8597844
- [Background] Hasegawa M, Kida S, Yamashima T, Yamashita J, Takakuwa S. Multicentric infantile myofibromatosis in the cranium: case report. Neurosurgery. 1995 Jun;36(6):1200-3. doi: 10.1227/00006123-199506000-00023. PMID 7644004
- [Background] Coffin CM, Dehner LP. Fibroblastic-myofibroblastic tumors in children and adolescents: a clinicopathologic study of 108 examples in 103 patients. Pediatr Pathol. 1991 Jul-Aug;11(4):569-88. doi: 10.3109/15513819109064791. PMID 1946077
- [Background] Stenzel P, Fitterer S. Gastrointestinal multicentric infantile myofibromatosis: characteristic histology on rectal biopsy. Am J Gastroenterol. 1989 Sep;84(9):1115-9. PMID 2672792
- [Background] Weyl Ben Arush M, Meller I, Moses M, Klausner J, Isakov J, Kuten A, el Hassid R. Multifocal desmoid tumor in childhood: report of two cases and review of the literature. Pediatr Hematol Oncol. 1998 Jan-Feb;15(1):55-61. doi: 10.3109/08880019809009508. PMID 9509506
- [Background] Riedlinger WF, Juraszek AL, Jenkins KJ, Nugent AW, Balasubramanian S, Calicchio ML, Kieran MW, Collins T. Pulmonary vein stenosis: expression of receptor tyrosine kinases by lesional cells. Cardiovasc Pathol. 2006 Mar-Apr;15(2):91-9. doi: 10.1016/j.carpath.2005.11.006. PMID 16533697
- [Background] Sadr IM, Tan PE, Kieran MW, Jenkins KJ. Mechanism of pulmonary vein stenosis in infants with normally connected veins. Am J Cardiol. 2000 Sep 1;86(5):577-9, A10. doi: 10.1016/s0002-9149(00)01022-5. PMID 11009286

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Avastin and/or Gleevec
Started | 50
Completed | 48
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Avastin and/or Gleevec
Number analyzed (Participants) | 48
Age, Customized [Count of Participants; unit: Participants]
  <3 months | 3
  3 to <6 months | 15
  6 to <12 months | 17
  >/= 12 months | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Survival at 48 Weeks
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Avastin and/or Gleevec: Patients were all treated with Gleevec (imatinib mesylate) and those without congenital heart disease, significant lung disease, and those who progressed were also treated with Avastin (bevacizumab).
Arm/Group | Avastin and/or Gleevec
Number analyzed (Participants) | 48
Participants | 42

2. Secondary Outcome: Number of Patients With Disease Progression at 48 Weeks
Description: Patients will be classified as having disease progression if at least 2 pulmonary veins have significantly worsened at 48 weeks. This determination is based on the study defined Pulmonary Vein Status Scale, which categorizes pulmonary veins on a scale from "1- None: No narrowing of the luminal contour," to "7- Distal atretic: Complete obliteration of the luminal contour extending >5mm within the vessel segment."
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Avastin and/or Gleevec
Number analyzed (Participants) | 48
Participants | 5

3. Secondary Outcome: Number of Patients With Disease Stabilization at 48 Weeks
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Avastin and/or Gleevec
Number analyzed (Participants) | 48
Participants | 15

ADVERSE EVENTS:
Arm/Group | Avastin and/or Gleevec
All-Cause Mortality (participants affected / at risk) | 11/48
Serious Adverse Events (participants affected / at risk) | 10/48
Other Adverse Events (participants affected / at risk) | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avastin and/or Gleevec (N=48)
Bone Marrow Suppression (Blood and lymphatic system disorders) | 2 (4)
Gastrointestinal Toxicity (Gastrointestinal disorders) | 4 (4)
Infection (Infections and infestations) | 5 (7)
Hospitalization (General disorders) | 2 (6)
Tremors (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avastin and/or Gleevec (N=48)
Blood Bone Marrow Suppression (Blood and lymphatic system disorders) | 48 (602)
Rash (Skin and subcutaneous tissue disorders) | 13 (16)
Gastrointestinal Toxicity (Gastrointestinal disorders) | 27 (65)
Infection (Infections and infestations) | 22 (50)
Liver Toxicity (General disorders) | 32 (127)
Renal Toxicity (Renal and urinary disorders) | 31 (184)
Transfusion (General disorders) | 6 (22)
Other (General disorders) | 41 (447)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No